CLINICAL TRIAL: NCT04961801
Title: Acalabrutinib for GVHD Prophylaxis in Allogeneic Hematopoietic Stem Cell Transplantation in Lymphomas and Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Manufacturer AstraZeneca withdrew the study due to lack of funding
Sponsor: Shin Mineishi (Other)
Collaborators: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor-Investigator, Shin Mineishi, Professor, Hematology/Oncology, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSCI-18-128
Record Dates: First submitted 2021-06-16; First posted 2021-07-14 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Lymphoma; Leukemia
Keywords: Graft-Versus-Host Disease Prophylaxis
MeSH Terms: conditions — Lymphoma; Leukemia | interventions — acalabrutinib; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib in combination with tacrolimus and methotrexate (Experimental): 1. Phase I: To determine the maximum tolerated dose (MTD) of Acalabrutinib in combination with tacrolimus and methotrexate for Phase II.
  2. Phase II: To determine if acalabrutinib in combination with tacrolimus and methotrexate is safe and effective in reducing acute GVHD rate.
  Interventions: Drug: Acalabrutinib, tacrolimus, methotrexate

INTERVENTIONS:
Drug: Acalabrutinib, tacrolimus, methotrexate — For Graft-Versus-Host Disease Prophylaxis in Allogeneic Hematopoietic Stem Cell Transplantation in Lymphomas and Leukemia

SUMMARY:
GVHD remains a major cause of morbidity and mortality following SCT. The current standard of care for prophylaxis against GVHD includes tacrolimus and methotrexate.

This study proposes to utilize acalabrutinib, a Bruton tyrosine kinase (BTK) inhibitor, for GVHD prophylaxis following allogeneic SCT.

The hypothesis is that the addition of acalabrutinib to our institutional standard GVHD prophylaxis (tacrolimus and methotrexate) is safe, feasible, and effective in reducing both the incidence and severity of acute GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to sign the study-specific informed consent form
2. Willingness to comply with all study procedures and attend all study visits.
3. Participant with (a) B-cell malignancies or (b) AML (CD117 positive) who are undergoing allogeneic SCT at Penn State Cancer Institute from an 8/8 matched unrelated donor. Donor selection and screening criteria are to comply with 21 CRF Part 1271.
4. Male or female participant, age ≥ 18 and ≤ 75 years.
5. Ability to swallow oral medication.
6. Women of childbearing potential (WOCP) as defined as not surgically sterile or not postmenopausal must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 7 days of beginning the condition regimen.
7. Men and WOCP must agree to use 2 medically accepted method of contraception and must agree to continue use this method while on the trial and through at least one week after the last dose of study drug. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD) known to have a failure rate of less than 1% per year, or steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) withdrawal, spermicides only, or lactational amenorrhea are not acceptable methods of contraception. WOCP must use a medically accepted method of contraception and must agree to continue use this method from the time of signing the informed consent through at least one week after the last dose of study drug.
8. Karnofsky Performance Scale (KPS) equal to or greater than 70%.

Exclusion Criteria:

1. Renal dysfunction with eGFR <30/mL/minute/1.73 m2 by Cockroft-Gault formula.
2. Participant requires warfarin or vitamin K antagonist within one week of acalabrutinib administration.
3. Participant requires treatment with a strong cytochrome P450 3A inducer or inhibitor.
4. Treatment with post-transplant cyclophosphamide
5. Treatment with any other investigational products within 21 days of conditioning regimen.
6. Known hypersensitivity to acalabrutinib, tacrolimus and methotrexate and their excipients.
7. Active uncontrolled infections
8. Human immunodeficiency virus (HIV) positivity.
9. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative polymerase chain reaction (PCR) and must be willing to undergo DNA PCR testing during the study to be eligible. Those who are HBsAg positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result to be eligible. Those who are hepatitis C PCR positive will be excluded.
10. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures.
11. Diagnosed or treated for another malignancy within 2 years before study registration or previously diagnosed with another malignancy and have any evidence of residual disease. Participant with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection.
12. Participant with coagulopathy or bleeding disorder.
13. Known hepatic cirrhosis or severe pre-existing hepatic impairment (ALT and/or AST more than 3x greater than upper limit of normal, Total Bilirubin more than 2x greater than upper limit of normal)
14. Uncontrolled high blood pressure (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg).
15. Uncontrolled or symptomatic cardiac arrhythmia
16. Left ventricular ejection fraction (LVEF) < 40% as assessed by echocardiogram or radionuclide angiography, or NYHA class 3 or 4 heart failure
17. Myocardial infarction within 6 months of signing consent.
18. History of stroke or intracranial hemorrhage within 6 months of signing consent.
19. Breastfeeding or pregnant.
20. Has difficulty with or is unable to swallow oral medication, or has significant gastrointestinal disease that would limit absorption of oral medication.
21. Suspected or confirmed PML(Progressive Multifocal Leukoencephalopathy)
22. Requires treatment with proton-pump inhibitors. (Participants receiving proton-pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment.)
23. FVC, FEV1, or DLCO (corrected with hemoglobin) less than 40% of expected value.
24. Prothrombin time (PT)/INR or aPTT (in the absence of lupus anticoagulant) >2x ULN.
25. Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
26. Concurrent participation in another therapeutic clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 30 days
  Dose-limiting toxicity of acalabrutinib in combination with tacrolimus and methotrexate in early SCT for Phase I part of the study
Maximum tolerated dose (MTD) | 30 days
  Maximum tolerated dose (MTD) of acalabrutinib in combination with tacrolimus and methotrexate in early SCT for Phase I part of the study
acute GVHD grade II-IV | 180 days
  Incidence of acute GVHD grade II-IV by day 180 for Phase II part of the study

IPD SHARING:
Plan to Share IPD: No